CLINICAL TRIAL: NCT07011147
Title: Primary Care Pragmatic, Real World Experience for Automated Insulin Delivery
Acronym: PREPARE 4 AID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Massachusetts General Hospital (Other); Beta Bionics, Inc. (Industry); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 24-0810; G-2312-06449 (Other Grant/Funding Number: The Leona M. and Harry B. Helmsley Charitable Trust)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes (T1D); Type 2 Diabetes; Diabetes, Autoimmune; Diabetes Mellitus; Diabetes Mellitus Type 2; Diabetes Mellitus, Type I; Diabetes, Type II; Diabetes; Diabetes Mellitus, Insulin-Dependent; Diabetes Mellitus Type II; Diabetes Type 2 on Insulin
Keywords: automated insulin delivery; type 1 diabetes; type 2 diabetes; bionic pancreas; closed loop; pancreas, artificial; t1d; t2d; diabetes; insulin; primary care
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: 13-week randomized controlled trial with optional 13-week extension phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bionic Pancreas (Experimental)
  Interventions: Device: Bionic Pancreas
- Routine Care (Active Comparator)
  Interventions: Other: Routine Care

INTERVENTIONS:
Device: Bionic Pancreas — The intervention group will use the iLet Bionic Pancreas (BP) for 13-weeks. They will be trained on the iLet BP system and its components by a Certified iLet Trainer. They will also be trained on how to use the study continuous glucose monitor (CGM) system, blood glucose meter, and ketone meter. Participants will have four mid-period follow up phone calls to review medications, ongoing eligibility, and solicit any occurrences of adverse events and device issues. At the end of 13-weeks, they will complete final visit tasks and will be transitioned back to their pre-study insulin delivery method with guidance provided by a study investigator.
  Arms: Bionic Pancreas
Other: Routine Care — Participants will continue with their current diabetes treatment. Participants will be trained on the use of the study blood glucose meter. They will have four mid-period follow up phone calls to review medications, ongoing eligibility, and solicit any occurrences of adverse events. At the end of 13-weeks, they will complete final visit tasks and will be asked if they would like to participate in the observational extension phase where they will use the iLet Bionic Pancreas for 13 weeks.
  Arms: Routine Care

SUMMARY:
The goal of this randomized controlled trial is to compare the efficacy and safety of the iLet Bionic Pancreas (BP) System in adults with insulin-treated diabetes (type 1 diabetes or type 2 diabetes) compared to standard of care when ordered by primary care providers. The main question it aims to answer is:

Can the iLet BP by deployed in primary care settings to adults with insulin-treated diabetes (type 1 diabetes or type 2 diabetes)?

Researchers will compare 13-weeks of iLet BP use to routine care to see if iLet BP use has a greater reduction in HbA1c compared to13-weeks of routine care.

Participants will:

Use the iLet BP for 13-weeks or continue their routine care Be trained to use the study devices or continue their routine care Complete a virtual screening visit, mid-period follow up calls and a final visit Complete baseline CGM collection Complete surveys and fingerstick a1c blood tests Routine care participants will have the option to complete an observational extension phase where they will wear the iLet BP for 13-weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent >18 and <89 years
2. Either 2.a. or 2.b.:

   1. Clinical diagnosis of type 1 diabetes for at least one year and using insulin for at least 1 year
   2. Clinical diagnosis of type 2 diabetes, on current injected or infused insulin regimen for at least 3 months prior to screening (e.g., basal-bolus, basal only, or pre-mix)
3. Stable doses of glucose lowering medications over the preceding 4 weeks as determined by Investigator, including GLP-1 receptor agonists (GLP-1 RA) and GLP-1/GIP RA agents
4. Stable doses of weight loss medications (including GLP-1 RA and GLP-1/GIP RA agents) over the preceding 4 weeks as determined by the investigator.
5. For those using the iLet Bionic Pancreas (during the RCT arm or observational extension phase), willingness to stay on current doses of medications throughout the study that may affect glycemia directly and/or indirectly, except for a dose reduction or discontinuation.
6. Have a primary care clinician willing to refer them to the study, confirm their diabetes diagnosis (for example: type 1 diabetes or type 2 diabetes), and recommend and manage the iLet for the duration of the study
7. Willing to comply with all study procedures for the duration of the study
8. Willing to wear a Dexcom CGM device and iLet system for duration of time randomized to iLet use or OEP
9. Willing to use the following insulin: lispro (including non-branded lispro and Humalog) or aspart (including non-branded aspart, Fiasp, and Novolog)
10. Investigator has confidence that the participant has the cognitive ability and can successfully operate all study devices and can adhere to the protocol
11. Willing and able to sign and date the Informed Consent Form (ICF)
12. If capable of becoming pregnant, willing and able to have pregnancy testing and use an acceptable method of contraception during the study period

    a. Capable of becoming pregnant means that menstruation has started and the participant is not surgically sterile or post-menopausal (12 months without menses) b. Acceptable methods of contraception include: i. Combined estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal).

    ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable).

    iii. Placement of an intrauterine device or intrauterine hormone-releasing system.

    iv. Barrier methods of contraception (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository).

    v. Has a vasectomized or sterile partner (where partner is sole partner of participant) and where vasectomy has been confirmed by medical assessment.

    vi. Exercises true sexual abstinence. Sexual abstinence is defined as refraining from heterosexual intercourse during the entire period of risk associated with the study.
13. Agreement to adhere to Lifestyle Considerations (see Section 5.3) throughout study duration
14. Have hardware and internet access capable of 2-way video and audio communication

Exclusion Criteria:

1. Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision or dexterity that prevents safe operation of the bionic pancreas, impaired memory)
2. Unable to speak and read English, as iLet BP support materials and device menus are currently available in English only
3. Diagnosis of maturity-onset diabetes of the young (MODY)
4. Plan to change usual diabetes regimen between screening and study randomization

   1. This would include changing from MDI to pump or from pump to MDI, starting a new class of type 2 diabetes medication, or starting or increasing GLP-1 RA or GLP-1/GIP RA medication
   2. This would NOT include changes to any insulin doses, including pump settings, short- and/or long-acting insulin doses and type of insulin; changing type 2 diabetes medication dosing (except GLP-1 RA or GLP-1/GIP RA); or changing type of type 2 diabetes medication within the same class
5. Weigh more than 255 kg (561 pounds) as this is the maximum weight that can be entered into the iLet user interface
6. History of bariatric surgery within 12 months prior to enrollment or plans for bariatric surgery within the period of study participation
7. Current use of a closed-loop or hybrid closed-loop insulin delivery system that is not FDA-cleared (e.g. "DIY Loop", "AAPS", "iAPS" or "Open APS")
8. Diagnosed blood disorder or dyscrasia associated with hemolysis, including for example: sickle cell disease and thalassemia, which in the Investigator's opinion could interfere with HbA1c accuracy
9. Planned use of hydroxyurea at any dose and/or of acetaminophen at doses exceeding 1 gram (1000 mg) every 6 hours.
10. Plans to receive a blood transfusion over the course of the study or has received a transfusion within 3 months prior to enrollment
11. Current participation in another diabetes-related clinical trial
12. History of diabetes due to cystic fibrosis, pancreatitis, or other pancreatic disease, including pancreatic tumor or insulinoma, or history of complete pancreatectomy
13. Have a history of intermittent oral or injectable glucocorticoid treatment within 8 weeks prior to screening or plans to take intermittent oral or injectable glucocorticoid during the study (chronic, stable treatment is acceptable, unplanned use is acceptable)
14. History of more than 1 episode of diabetic ketoacidosis (DKA) or hyperglycemic hyperosmolar syndrome (HHS) in the 6 months prior to screening, unrelated to an intercurrent illness or to a kinked, dislodged, or occluded cannula
15. Established history of allergy or severe reaction to adhesive or tape that must be used in the study
16. Treated currently or within the past 30 days prior to enrollment, or plan to begin treatment, with sulfonylurea, pramlintide, or SGLT-2 inhibitor medication
17. Any planned surgery during the study that would be considered major in the opinion of the investigator
18. Pregnant or lactating, or planning to become pregnant in the next 6 months
19. Renal failure on dialysis or chronic renal disease with a GFR or eGFR <30mL/min (values within the last two years will be accepted; if none available or >2 years prior, participant will be instructed to obtain GFR or eGFR through their usual care provider and to make copy of result available to study team)
20. Any condition or circumstance that, in the opinion of the site principal investigator, could interfere with the safe or effective completion of the study or which could compromise the results of the study c. Conditions to be considered by the investigator may include, but are not limited to, the following: i. Active clinical diagnosis of substance use disorder ii. Chronic use of opiates and/or benzodiazepines which, in the opinion of the investigator, might make it difficult for the participant to follow study procedures iii. Coronary artery disease that is not stable with medical management, including unstable angina, angina that prevents moderate exercise (e.g. exercise of intensity up to 6 METS) despite medical management, or within the last 12 months before screening, a history of myocardial infarction, percutaneous coronary intervention, enzymatic lysis of a presumed coronary occlusion, or coronary artery bypass grafting iv. Known history of prolonged QTc interval, malignant arrhythmia, or severe congenital heart disease v. Congestive heart failure with New York Heart Association (NYHA) Functional Classification III or IV vi. History of TIA or stroke in the last 12 months vii. Untreated or inadequately treated mental illness viii. History of untreated or inadequately treated eating disorder within the last 2 years, such as anorexia, bulimia, or diabulimia, or omission of insulin to manipulate weight ix. History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
21. Plans to travel outside of the US and its territories for more than four weeks consecutively
22. Plans not to have internet/video/phone access for more than one week consecutively
23. Employed by, or having immediate family members employed by Beta Bionics, or being directly involved in conducting the clinical trial, or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial
24. Previous use of the iLet for more than four weeks (including use of the commercially available iLet or prior participation in a study involving wearing the iLet for more than four weeks)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c between the BP and RC groups | RCT Week 13
  Superiority testing for HbA1c at 13 weeks between the BP and RC groups using linear mixed effects regression models adjusting for baseline HbA1c.
Percentage of Time With CGM Glucose <54 mg/dl | RCT Weeks 1-13 and OEP Weeks 13-26
  Non-inferiority testing for ordinal TBR<54mg/dL will be determined using a two-sided 95% confidence interval on the mean difference in % time <54 mg/dL between BP and RC groups using a linear mixed effects regression model adjusting for baseline % time <54 mg/dL, diabetes type, and clinical center.

SECONDARY OUTCOMES:
Percentage of Time With CGM Glucose in the 70-180 mg/dl Range | RCT Weeks 1-13 and OEP Weeks 13-26
  Calculated from all individual CGM values from RCT weeks 1-13 for each participant.
Percentage of Time in Tight Range With CGM Glucose in the 70-140 mg/dl | RCT Weeks 1-13 and OEP Weeks 13-26
  Calculated from all individual CGM values from weeks 1-13 for each participant.
Mean CGM Glucose | RCT Weeks 1-13 and OEP Weeks 13-26
  Individual CGM values from weeks 1-13 averaged together for each participant.
Percentage of Time With CGM Glucose >250 mg/dl Range | RCT Weeks 1-13 and OEP Weeks 13-26
  Calculated from all individual CGM values from weeks 1-13 for each participant.
Percentage of Time With CGM Glucose >180 mg/dl Range | RCT Weeks 1-13 and OEP Weeks 13-26
  Calculated from all individual CGM values from weeks 1-13 for each participant.
Standard deviation of CGM glucose | RCT Weeks 1-13 and OEP Weeks 13-26
  Calculated from mean CGM values from weeks 1-13 for each participant.
Percentage of Time With CGM Glucose Below <70 mg/dl Range | RCT Weeks 1-13 and OEP Weeks 13-26
  Calculated from all individual CGM values from weeks 1-13 for each participant.
Percentage of Time With CGM Glucose Below <54 mg/dl Range | RCT Weeks 1-13 and OEP Weeks 13-26
  Calculated from all individual CGM values from weeks 1-13 for each participant.
Coefficient of variation of CGM glucose | RCT Weeks 1-13 and OEP Weeks 13-26
  Calculated from mean CGM values from weeks 1-13 for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Oser, MD, MPH, CDCES, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Deidentified glucose data and psychosocial data will be shared with research collaborators.
Supporting Information: Study Protocol